CLINICAL TRIAL: NCT02811263
Title: High-dose Erythropoietin for Asphyxia and Encephalopathy
Acronym: HEAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other); Pediatrix (Other); University of Utah (Other); Children's National Research Institute (Other); University of Minnesota (Other); University of Texas (Other); Washington University School of Medicine (Other); Indiana University (Other); Stanford University (Other); University of Pittsburgh (Other); Children's Hospital Los Angeles (Other); Nationwide Children's Hospital (Other); Boston University (Other); University of New Mexico (Other); University of Chicago (Other); University of North Carolina (Other); Vanderbilt University (Other); Children's Hospital Medical Center, Cincinnati (Other); Johns Hopkins University (Other); Cook Children's Medical Center (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Yvonne Wu, Professor of Neurology and Pediatrics, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0511976
Record Dates: First submitted 2016-06-17; First posted 2016-06-23 (Estimated); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Neonatal Encephalopathy; Birth Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Active Comparator): Erythropoietin 1000 U/kg IV, at about 1, 2, 3, 4, and 7 days of age (i.e., 5 doses)
  Interventions: Drug: Erythropoietin
- Placebo (Placebo Comparator): Normal saline IV (equal volume), at about 1, 2, 3, 4, and 7 days of age
  Interventions: Drug: Normal saline placebo

INTERVENTIONS:
Drug: Normal saline placebo — Equal volume of normal saline to be used as placebo
  Other Names: NS
  Arms: Placebo
Drug: Erythropoietin — Epogen drawn from commercially available single dose 4000U/mL vials
  Other Names: Epogen
  Arms: Erythropoietin

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) occurs when a baby gets reduced blood flow and oxygen to the brain near the time of birth. This results in death or neurologic disabilities including cerebral palsy and cognitive impairment in up to half of affected infants. This clinical trial will determine if the drug erythropoietin (Epo) added to hypothermia (usual therapy) will improve outcomes for infants suffering from HIE.

DETAILED DESCRIPTION:
Neonatal hypoxic-ischemic encephalopathy (HIE) refers to brain injury resulting from reduced blood and oxygen flow to a baby's brain near the time of birth. HIE affects up to 12,000 newborns each year in the U.S. Half of affected infants have a bad outcome including death, cerebral palsy and cognitive impairment despite receiving hypothermia, the only available treatment. Erythropoietin (Epo) is a cytokine with remarkable neuroprotective and neuroregenerative effects demonstrated in animal models of neonatal brain injury. In a phase I trial of Epo + hypothermia, the investigators found that Epo 1000 U/Kg/dose best reproduced the pharmacokinetics of neuroprotective dosing in animal models. Long term outcomes were better than expected based on entry criteria and MRI findings. A phase II trial compared 50 cooled infants randomized to receive Epo or placebo. Infants treated with hypothermia + Epo had less brain injury on early MRI, and better 12-month motor development. The investigators hypothesize that Epo given to cooled infants with moderate/severe HIE will reduce the combined primary outcome of death or neurodevelopmental impairment from 49 to 33%. This is a randomized, double-blind, placebo-controlled trial of Epo therapy in 500 infants with HIE undergoing hypothermia. Specific aims are 1) To determine if 5 doses of Epo 1000 U/kg IV reduces the rate of death, motor or cognitive deficits at 2 years; 2) To assess safety of Epo by evaluating clinical toxicity; and 3) To determine whether Epo decreases the severity of neonatal brain injury as evidenced by early MRI and circulating biomarkers of brain injury. The investigators anticipate that Epo will confer improved 2-year neurodevelopmental outcome, will be safe, and will decrease brain injury severity as determined by early biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 36 weeks of gestational age
* Receiving active or passive whole body cooling/hypothermia since < 6 hours of age
* Perinatal depression based on at least one of the following:

  1. Apgar score < 5 at 10 minutes, or
  2. Need for resuscitation at 10 minutes (i.e., chest compressions, or positive pressure respiratory support including endotracheal, mask ventilation, or CPAP), or
  3. pH < 7.00 in cord gas (arterial or venous) or in an infant gas (arterial or venous) obtained at < 60 minutes of age, or
  4. Base deficit ≥ 15 mmol/L in cord gas (arterial or venous) or in an infant gas (arterial or venous) obtained at < 60 minutes of age
* Moderate to severe encephalopathy (based on modified Sarnat exam) present between 1-6 hours after birth

Exclusion Criteria:

* Study drug unlikely to be administered within 26 hours of birth
* Infant has living twin (or higher order multiple) who is also being cooled
* Birth weight < 1800 g (e.g., intrauterine growth restriction)
* Genetic or congenital condition that affects neurodevelopment or requires multiple surgeries (e.g., congenital viral infection, hydrops, complex congenital heart disease, severe dysmorphic features, etc.)
* Head circumference < 30 cm
* Redirection of care is being considered due to moribund condition
* Patient anticipated to be unavailable for evaluation at age 2
* Polycythemia (hematocrit > 65.0%)
* Parents/legal guardians with diminished capacity and autonomy
* Infant is participating or intends to participate in another interventional study during the birth hospitalization (note: does not include observational studies)
* Sentinel event and encephalopathy occurred only after birth
* Unable to consent in primary language of parent(s)

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Wu, MD MPH, Principal Investigator — University of California, San Francisco; Sandra Juul, MD PHD, Principal Investigator — University of Washington
Locations (23):
- United States (23):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Children's Hospitals and Clinics of Minnesota: Minneapolis, Minneapolis, Minnesota
  - Children's Hospitals and Clinics of Minnesota: St. Paul, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Juul SE, Comstock BA, Heagerty PJ, Mayock DE, Goodman AM, Hauge S, Gonzalez F, Wu YW. High-Dose Erythropoietin for Asphyxia and Encephalopathy (HEAL): A Randomized Controlled Trial - Background, Aims, and Study Protocol. Neonatology. 2018;113(4):331-338. doi: 10.1159/000486820. Epub 2018 Mar 7. PMID 29514165
- [Background] Wisnowski JL, Bluml S, Panigrahy A, Mathur AM, Berman J, Chen PK, Dix J, Flynn T, Fricke S, Friedman SD, Head HW, Ho CY, Kline-Fath B, Oveson M, Patterson R, Pruthi S, Rollins N, Ramos YM, Rampton J, Rusin J, Shaw DW, Smith M, Tkach J, Vasanawala S, Vossough A, Whitehead MT, Xu D, Yeom K, Comstock B, Heagerty PJ, Juul SE, Wu YW, McKinstry RC; HEAL Study Group. Integrating neuroimaging biomarkers into the multicentre, high-dose erythropoietin for asphyxia and encephalopathy (HEAL) trial: rationale, protocol and harmonisation. BMJ Open. 2021 Apr 22;11(4):e043852. doi: 10.1136/bmjopen-2020-043852. PMID 33888528
- [Result] Chalak L, Redline RW, Goodman AM, Juul SE, Chang T, Yanowitz TD, Maitre N, Mayock DE, Lampland AL, Bendel-Stenzel E, Riley D, Mathur AM, Rao R, Van Meurs KP, Wu TW, Gonzalez FF, Flibotte J, Mietzsch U, Sokol GM, Ahmad KA, Baserga M, Weitkamp JH, Poindexter BB, Comstock BA, Wu YW. Acute and Chronic Placental Abnormalities in a Multicenter Cohort of Newborn Infants with Hypoxic-Ischemic Encephalopathy. J Pediatr. 2021 Oct;237:190-196. doi: 10.1016/j.jpeds.2021.06.023. Epub 2021 Jun 16. PMID 34144032
- [Result] Wu YW, Comstock BA, Gonzalez FF, Mayock DE, Goodman AM, Maitre NL, Chang T, Van Meurs KP, Lampland AL, Bendel-Stenzel E, Mathur AM, Wu TW, Riley D, Mietzsch U, Chalak L, Flibotte J, Weitkamp JH, Ahmad KA, Yanowitz TD, Baserga M, Poindexter BB, Rogers EE, Lowe JR, Kuban KCK, O'Shea TM, Wisnowski JL, McKinstry RC, Bluml S, Bonifacio S, Benninger KL, Rao R, Smyser CD, Sokol GM, Merhar S, Schreiber MD, Glass HC, Heagerty PJ, Juul SE; HEAL Consortium. Trial of Erythropoietin for Hypoxic-Ischemic Encephalopathy in Newborns. N Engl J Med. 2022 Jul 14;387(2):148-159. doi: 10.1056/NEJMoa2119660. PMID 35830641
- [Derived] Lew CO, Calabrese E, Chen JV, Tang F, Chaudhari G, Lee A, Faro J, Juul S, Mathur A, McKinstry RC, Wisnowski JL, Rauschecker A, Wu YW, Li Y. Artificial Intelligence Outcome Prediction in Neonates with Encephalopathy (AI-OPiNE). Radiol Artif Intell. 2024 Sep;6(5):e240076. doi: 10.1148/ryai.240076. PMID 38984984
- [Derived] Rao R, Comstock BA, Wu TW, Mietzsch U, Mayock DE, Gonzalez FF, Wood TR, Heagerty PJ, Juul SE, Wu YW. Time to Reaching Target Cooling Temperature and 2-year Outcomes in Infants with Hypoxic-Ischemic Encephalopathy. J Pediatr. 2024 Mar;266:113853. doi: 10.1016/j.jpeds.2023.113853. Epub 2023 Nov 23. PMID 38006967
- [Derived] Gonzalez FF, Voldal E, Comstock BA, Mayock DE, Goodman AM, Cornet MC, Wu TW, Redline RW, Heagerty P, Juul SE, Wu YW. Placental Histologic Abnormalities and 2-Year Outcomes in Neonatal Hypoxic-Ischemic Encephalopathy. Neonatology. 2023;120(6):760-767. doi: 10.1159/000533652. Epub 2023 Sep 22. PMID 37742617
- [Derived] Calabrese E, Wu Y, Scheffler AW, Wisnowski JL, McKinstry RC, Mathur A, Glass HC, Comstock BA, Heagerty PJ, Gillon S, Juul SE, Hess CP, Li Y. Correlating Quantitative MRI-based Apparent Diffusion Coefficient Metrics with 24-month Neurodevelopmental Outcomes in Neonates from the HEAL Trial. Radiology. 2023 Sep;308(3):e223262. doi: 10.1148/radiol.223262. PMID 37698478
- [Derived] Juul SE, Voldal E, Comstock BA, Massaro AN, Bammler TK, Mayock DE, Heagerty PJ, Wu YW, Numis AL; HEAL consortium. Association of High-Dose Erythropoietin With Circulating Biomarkers and Neurodevelopmental Outcomes Among Neonates With Hypoxic Ischemic Encephalopathy: A Secondary Analysis of the HEAL Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2322131. doi: 10.1001/jamanetworkopen.2023.22131. PMID 37418263
- [Derived] Juul SE, Comstock BA, Cornet MC, Gonzalez FF, Mayock DE, Glass HC, Schreiber MD, Heagerty PJ, Wu YW. Safety of High Dose Erythropoietin Used with Therapeutic Hypothermia as Treatment for Newborn Hypoxic-Ischemic Encephalopathy: Secondary Analysis of the HEAL Randomized Controlled Trial. J Pediatr. 2023 Jul;258:113400. doi: 10.1016/j.jpeds.2023.113400. Epub 2023 Apr 4. PMID 37019334

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erythropoietin | Placebo
Started | 257 | 243
Completed | 240 | 222
Not Completed | 17 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin | Placebo | Total
Number analyzed (Participants) | 257 | 243 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (6.3) | 30.0 (6.6) | 29.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 103 | 225
  Male | 135 | 140 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 59 | 122
  Not Hispanic or Latino | 194 | 184 | 378
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 15 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 38 | 66
  White | 183 | 173 | 356
  More than one race | 10 | 6 | 16
  Unknown or Not Reported | 18 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States | 257 | 243 | 500
Maternal education, high school or less [Count of Participants; unit: Participants] | 102 | 83 | 185
Parity of 1, including trial infant [Count of Participants; unit: Participants] | 145 | 141 | 286
Pregnancy and delivery complications - maternal chorioamnionitis or fever [Count of Participants; unit: Participants] | 45 | 32 | 77
Pregnancy and delivery complications - maternal preeclampsia or eclampsia [Count of Participants; unit: Participants] | 22 | 23 | 45
Pregnancy and delivery complications - gestational diabetes [Count of Participants; unit: Participants] | 33 | 25 | 58
Pregnancy and delivery complications - maternal obesity: body-mass index >30 [Count of Participants; unit: Participants] | 47 | 42 | 89
Pregnancy and delivery complications - sentinel event [Count of Participants; unit: Participants] | 71 | 72 | 143
Pregnancy and delivery complications - sentinel event (shoulder dystocia) [Count of Participants; unit: Participants] | 14 | 18 | 32
Pregnancy and delivery complications - sentinel event (placental abruption) [Count of Participants; unit: Participants] | 40 | 31 | 71
Pregnancy and delivery complications - sentinel event (prolapsed cord) [Count of Participants; unit: Participants] | 10 | 13 | 23
Pregnancy and delivery complications - sentinel event (uterine rupture) [Count of Participants; unit: Participants] | 13 | 11 | 24
Pregnancy and delivery complications - Cesarean section delivery [Count of Participants; unit: Participants] | 170 | 159 | 329
Pregnancy and delivery complications - outborn delivery [Count of Participants; unit: Participants] | 214 | 201 | 415
Infant birth weight [Mean (Standard Deviation); unit: grams] | 3332 (572) | 3414 (614) | 3372 (594)
Infant gestational age [Mean (Standard Deviation); unit: weeks] | 39.1 (1.4) | 39.2 (1.5) | 39.1 (1.5)
Infant 5-minute Apgar score [Median (Inter-Quartile Range); unit: score on a scale] — The Apgar score is a calculated score, with 10 being the maximum score. An infant receives a score of 0, 1, or 2 for each of the following: heart rate, breathing, color, activity, grimace. These sub-scores are added together, and the higher the score, the better the infant appears. This evaluation is typically done at 1, 5, and 10 minutes after birth.
  score on a scale | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 5]
Infant 10-minute Apgar score [Median (Inter-Quartile Range); unit: score on a scale] — The Apgar score is a calculated score, with 10 being the maximum score. An infant receives a score of 0, 1, or 2 for each of the following: heart rate, breathing, color, activity, grimace. These sub-scores are added together, and the higher the score, the better the infant appears. This evaluation is typically done at 1, 5, and 10 minutes after birth.
  score on a scale | 5 [3 to 7] | 5 [3.8 to 6] | 5 [3 to 7]
Infant - continued resuscitation at 10 minutes [Count of Participants; unit: Participants] | 243 | 217 | 460
Infant - lowest pH [Mean (Standard Deviation); unit: pH] | 6.95 (0.17) | 6.91 (0.17) | 6.93 (0.17)
Infant - severe encephalopathy [Count of Participants; unit: Participants] — Enrolled infants had either moderate or severe encephalopathy, based on the presence of at least 3 of 6 Sarnat criteria present between 1-6 hours after birth. The HEAL study used a modified Sarnat scoring system that assessed: level of consciousness, spontaneous activity, posture, tone, primitive reflexes (suck and moro), and autonomic (pupils and respiration).
  Participants | 59 | 54 | 113
Infant - age at randomization [Median (Inter-Quartile Range); unit: hours] | 14 [10 to 19] | 14 [10 to 20] | 14 [10 to 20]
Infant - age at first treatment [Mean (Standard Deviation); unit: hours] | 17.6 (5.5) | 17.6 (5.5) | 17.6 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or Neurodevelopmental Impairment
Description: Neurodevelopmental impairment defined as any of the following: a) Gross Motor Function Scale (GMFCS) level ≥ 1, or b) GMFCS = 0 or 0.5 and cerebral palsy (CP) (any type), or c) Bayley III Cognitive Score < 90
Time Frame: Prior to final outcome assessment at 22-26 months of age; For extenuating circumstances, for example, COVID-19 restrictions, may be performed up to 36 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 240 | 222
Participants | 126 | 110

2. Secondary Outcome: Number of Participants With Cerebral Palsy (CP) and Number of Participants With Each Type of Cerebral Palsy (CP), Determined Using a Standardized Neurologic Examination
Description: Neurologic diagnoses: no CP, diparetic CP, hemiparetic CP, quadriparetic CP
Time Frame: 22-26 months; For extenuating circumstances, for example, COVID-19 restrictions, may be performed up to 36 months of age
Population: All toddlers evaluated with a neuro exam at 22-26 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 207 | 198
Participants
  No cerebral palsy | 176 | 173
  Diparetic cerebral palsy | 9 | 6
  Hemiparetic cerebral palsy | 3 | 2
  Quadriparetic cerebral palsy | 19 | 17

3. Secondary Outcome: Number of Participants With Each Level of Gross Motor Function, Determined Using the GMFCS
Description: Gross Motor Function Scale (GMFCS) is a scale from 0-5, with higher values representing worse outcomes.
  * Level 0: Walks 10 steps independently with symmetrical gait
  * Level 0.5: Walks 10 steps independently without symmetrical gait
  * Level 1: Sits. Hands free for play, and creeps or crawls on hands and knees, pulls to stand; cruises or walks with hands held
  * Level 2: Uses hands for sitting support; creeps on stomach or crawls, may cruise/pull to stand
  * Level 3: Sits with external support for lower trunk; rolls, creeps on stomach
  * Level 4: Good head control in supported sitting; can roll to supine, may roll to prone
  * Level 5: Unable to maintain anti-gravity head and trunk postures in prone or sitting; little or no voluntary movement.
Time Frame: as for outcome 2
Population: The analysis population includes participants with GMFCS score available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) is higher, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 211 | 204
Participants
  GMFCS = 0 | 186 | 178
  GMFCS = 0.5 | 6 | 6
  GMFCS = 1 | 4 | 6
  GMFCS = 2 | 3 | 5
  GMFCS = 3 | 2 | 1
  GMFCS = 4 | 4 | 1
  GMFCS = 5 | 6 | 7

4. Secondary Outcome: Bayley III Cognitive Score
Description: The Bayley III cognitive score is a population normed score. 100 indicates the population mean with a standard deviation of 15; higher scores indicate a higher level of development.
Time Frame: as for outcome 2
Population: The analysis population includes participants with Bayley III cognitive score available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) is higher, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 200 | 192
score on a scale | 89.1 (15.7) | 89.5 (17.5)

5. Secondary Outcome: Bayley III Language Score
Description: The Bayley III language score is a population normed score. 100 indicates the population mean with a standard deviation of 15; higher scores indicate a higher level of development.
Time Frame: as for outcome 2
Population: The analysis population includes participants with Bayley III language score available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) is higher, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 198 | 188
score on a scale | 87.9 (20.4) | 86.7 (20.8)

6. Secondary Outcome: Number of Participants With Epilepsy
Description: ≥ 2 afebrile, unprovoked seizures
Time Frame: Prior to 22-26 months
Population: The analysis population includes participants with data regarding epilepsy available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) is higher, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Count of Participants; unit: Participants
Groups:
- Erythropoietin: Erythropoietin treated.
- Placebo: Placebo treated.
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 210 | 205
Participants | 5 | 4

7. Secondary Outcome: Number of Participants With Behavioral Abnormalities Determined by the Externalizing Score of the Child Behavior Checklist
Description: Score for externalizing problems on Childhood Behavior Checklist of >= 65
Time Frame: 22-26 months
Population: The analysis population includes participants with Child Behavior Checklist scores available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) is higher, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 207 | 201
Participants | 15 | 3

8. Other Pre Specified Outcome: Number of Participants at Each Level of Severity of Impairment [(1) Normal, (2) Mild Motor and/or Cognitive Impairment, (3) Moderate/Severe Motor and or Cognitive Impairment, (4) Death], Compared Between the Epo and Placebo Groups.
Description: Mild impairment: GMFCS=1 and no cerebral palsy, or GMFCS<=0.5 and hemiplegic or diplegic cerebral palsy.
  Moderate/severe impairment: GMFCS=1 and cerebral palsy, GMFCS >=2, quadriplegic cerebral palsy, or Bayley III cognitive score <85.
Time Frame: Through 22-26 months
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 240 | 222
Participants
  Normal | 114 | 112
  Mild motor and/or cognitive impairment | 26 | 23
  Moderate/severe impairment | 63 | 59
  Death | 37 | 28

9. Other Pre Specified Outcome: Rates of Epo-related Adverse Events
Time Frame: Through hospital discharge
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Rates of Epo-related Adverse Events
Time Frame: Through 22-26 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Serial Circulating Biomarkers of Inflammation/Brain Injury
Description: Epo level at baseline, day 2, and day 4.
Time Frame: During first week of life
Population: The analysis population includes participants with biologic samples available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) differs, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Median (Inter-Quartile Range); unit: mU/ml
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 228 | 217
mU/ml
  Baseline | 32.7 [13.5 to 183.4] | 36.0 [12.3 to 96.7]
  Day 2 | 1530 [1259 to 5802] | 34.4 [18.0 to 91.9]
  Day 4 | 2682 [2190 to 4637] | 20.5 [8.1 to 54.7]

12. Other Pre Specified Outcome: MR Evidence of Brain Injury - Brain Injury Score
Description: Global brain injury scores were calculated using a validated scoring system for HIE. The extent of injury was recorded (i.e., none = 0, <25% = 1, 25-50% = 2; >50% = 3) as seen on T1, T2, and apparent diffusion coefficient (ADC) images in 8 regions of the brain: caudate, putamen/globus pallidus, thalamus, posterior limb of t he internal capsule (PLIC), cortex, white matter, brainstem, and cerebellum. The severity of brain injury was determined from the global injury score as follows: none (global injury score = 0), mild (1-11), moderate (12-32), or severe (33-138).
Time Frame: During first week of life
Population: The analysis population includes participants with brain MRI data from the first week of life available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) differs, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 242 | 231
score on a scale | 8 [2 to 26] | 7 [2 to 20]

13. Other Pre Specified Outcome: Number of Participants With MR Evidence of Brain Injury - Severity of Brain Injury
Time Frame: During first week of life
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 242 | 231
Participants
  None | 49 | 51
  Mild | 91 | 86
  Moderate | 46 | 51
  Severe | 56 | 43

14. Other Pre Specified Outcome: Number of Participants Experiencing Hearing Impairment Requiring Hearing Aids, Per Parent/Caregiver Report, Compared Between the Epo and Placebo Groups.
Time Frame: Through 22-26 months
Population: The analysis population includes participants with hearing impairment data available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) differs, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 211 | 203
Participants | 10 | 13

15. Other Pre Specified Outcome: Number of Participants Experiencing Cortical Visual Impairment, Per Parent/Caregiver Report, Compared Between the Epo and Placebo Groups.
Time Frame: Through 22-26 months
Population: The analysis population includes participants with visual impairment data available. Total number of participants analyzed in the Participant Flow module (N=240, N=222) differs, as it reflects participants for whom the primary endpoint of death or neurodevelopmental impairment (NDI) could be determined. The primary endpoint can be determined when thresholds are met on either neurologic examination, Bayley III cognitive score, or GMFCS score, or when death occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Erythropoietin | Placebo
Number analyzed (Participants) | 211 | 203
Participants | 19 | 20

ADVERSE EVENTS:
Time Frame: Adverse Events were collected through hospital discharge from birth, regardless of duration of hospitalization (mean = 21.4 days; median = 14 days; range = 5-187 days). Serious Adverse Events were collected through 30 days of study drug dosing. Death occurring at any time during the neonatal or follow-up period (up to 36 months) was also reported as a Serious Adverse Event.
Description: Adverse Events: anticipated medical complications of hypoxic-ischemic encephalopathy.
  Serious Adverse Events: systemic hypertension, polycythemia, disseminated intravascular coagulation, major venous or arterial thrombosis (clot), pulmonary hypertension, intracranial hemorrhage, cardiopulmonary arrest, other unexpected life-threatening event, death.
Arm/Group | Erythropoietin | Placebo
All-Cause Mortality (participants affected / at risk) | 37/257 | 28/243
Serious Adverse Events (participants affected / at risk) | 137/257 | 106/243
Other Adverse Events (participants affected / at risk) | 254/257 | 240/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoietin (N=257) | Placebo (N=243)
Death (General disorders) | 37 | 28
Systemic hypertension (Cardiac disorders) | 7 | 7 — Blood pressure elevated enough to require antihypertensive therapy
Polycythemia (Blood and lymphatic system disorders) | 0 | 0 — Central hematocrit (Hct) > 65.0%, as measured by a central lab on 2 consecutive free-flowing arterial or venous samples.
Major venous or arterial thrombosis (Blood and lymphatic system disorders) | 6 | 3 — Any thrombosis treated with course of anticoagulation. Any venous or arterial thrombosis involving major vessel not related to a central line. Any symptomatic thrombosis involving major vessel (e.g., symptoms such as superior vena cava syndrome).
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 39 | 25 — Clinical bleeding or oozing requiring transfusion of blood products (e.g., fresh frozen plasma, cryoprecipitate, or platelets).
Pulmonary hypertension (Cardiac disorders) | 51 | 36 — Elevated pulmonary vascular resistance treated with inhaled nitric oxide or extracorporeal membrane oxygenation (ECMO) therapy
Intracranial hemorrhage (Blood and lymphatic system disorders) | 68 | 55 — Intraparenchymal or intraventricular blood visualized by head ultrasound or MRI T1 or T2 sequences.
Cardiopulmonary arrest (Cardiac disorders) | 3 | 3 — Clinical code event requiring chest compressions or epinephrine bolus from which the infant recovers (does not lead to death), that is not secondary to endotracheal tube obstruction or other mechanical issue.
Other unexpected life threatening event (General disorders) | 10 | 6 — Unexpected for hypoxic-ischemic encephalopathy, or unexpected based on the erythropoietin drug profile.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erythropoietin (N=257) | Placebo (N=243)
Intubated > 7 days (Respiratory, thoracic and mediastinal disorders) | 49 | 38
Ever intubated (Respiratory, thoracic and mediastinal disorders) | 206 | 195
Meconium aspiration system (Respiratory, thoracic and mediastinal disorders) | 46 | 49
Hypotension warranting inotropes (Cardiac disorders) | 90 | 73
Dysrhythmia (Cardiac disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 115 | 88
Neutropenia (Blood and lymphatic system disorders) | 24 | 17
Acute kidney injury (Renal and urinary disorders) | 35 | 23
Acute liver injury (Hepatobiliary disorders) | 125 | 111
Seizure: clinical or electrographic (Nervous system disorders) | 88 | 97
Discharged alive - abnormal neurologic examination (Nervous system disorders) | 50 | 58
Discharged alive - nasal cannula oxygen (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Discharged alive - tracheostomy or ventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Discharged alive - nasogastric tube feeding (Gastrointestinal disorders) | 5 | 3
Discharged alive - gastrostomy tube feeding (Gastrointestinal disorders) | 17 | 19
Discharged alive - failed hearing screening (Ear and labyrinth disorders) | 17 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02811263/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT02811263/SAP_001.pdf